CLINICAL TRIAL: NCT01518478
Title: An Open Label Study in Adults With Atopic Dermatitis to Assess Variability in Immune Response to Fluzone® Intradermal Vaccine
Brief Title: Atopic Dermatitis Research Network (ADRN) Influenza Vaccine Pilot
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Atopic Dermatitis Research Network (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DAIT ADRN-03
Record Dates: First submitted 2011-12-14; First posted 2012-01-26 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 20 Non-atopic (Other): Non-atopic, healthy control.
  Interventions: Drug: Fluzone® Intradermal (Sanofi Pasteur Inc.)
- 20 ADEH- (mild to severe AD) (Other): Atopic Dermatitis without previous or current Eczema Herpeticum.
  Interventions: Drug: Fluzone® Intradermal (Sanofi Pasteur Inc.)

INTERVENTIONS:
Drug: Fluzone® Intradermal (Sanofi Pasteur Inc.) — Fluzone® Intradermal trivalent vaccine is a clear-to-slightly opalescent, preservative-free suspension containing formaldehyde-inactivated "split" influenza viruses for intradermal delivery of 0.1 mL via an ultra-fine micro-needle. The vaccine is supplied as a single-dose, in a latex-free, pre-filled microinjection system. The active substance is prepared from influenza viruses propagated in embryonated chicken eggs.
  Fluzone® Intradermal is standardized according to United States Public Health Service (US PHS) requirements and is formulated to contain HA of each of the following three influenza strains recommended for the 2011-2012 influenza season: A/California/07/2009 X-179A (H1N1)-like virus, A/Perth/16/2009 (H3N2)-like virus, and B/Brisbane/60/2008-like virus.

SUMMARY:
A new flu vaccine which is injected into the skin instead of into the muscle has recently been approved by the Food and Drug Administration for vaccination of the general population including patients with atopic dermatitis (AD). This new vaccine has been shown to work as well as the vaccine which is injected into muscle when tested in people without atopic dermatitis. The primary endpoint of the study is to estimate the variance of the log fold change from baseline in HAI antibody titers for non-atopic controls and participants with atopic dermatitis without a history of eczema herpeticum (ADEH-), following administration of a single dose of the seasonal 2011-2012 Fluzone® Intradermal vaccine.

DETAILED DESCRIPTION:
This is a single center, open-label, mechanistic study designed to determine the variance of the antibody response in non-atopic and ADEH- participants receiving a single dose of the 2011-2012 seasonal Fluzone® Intradermal vaccine administered per label.

Twenty non-atopic and 20 ADEH- (mild to severe AD) adults aged 18 to 64 years will be enrolled. Enrollment will be closely monitored to ensure that there is a similar distribution of non-atopic and ADEH- participants by gender, age, and race/ethnicity.

Eligible study participants will provide a pre-vaccination blood sample (Day 0) for assessment of baseline HAI antibody titers, cellular immune response, total IgE, and allergen sensitization, and will then receive a single injection of the 2011-2012 seasonal Fluzone® Intradermal vaccine administered per label. A subset of participants will also provide blood for microarray analysis at Baseline (Day 0) and will return to the clinic 3 and 7 days post-vaccination to provide additional blood for microarray analysis. All participants will return to the study site 28 days post-vaccination for a blood draw for HAI antibody titers and cellular immune response assays.

Study participants will be followed for safety, including serious adverse events (SAEs), throughout the entire duration of the study and will be asked to record solicited AEs on a diary card (Days 0-7).

ELIGIBILITY:
Inclusion Criteria:

Participants who meet all of the following criteria are eligible for enrollment.

* Who are males and females 18 to 64 years of age, inclusive, on the day of vaccination.
* Who are enrolled in the ADRN Registry study.
* Who have active, mild to severe AD without a history of EH or who are non-atopic as diagnosed using the ADRN Standard Diagnostic Criteria. Non-atopic status will be based on self-reported history and will not take total IgE or allergen sensitization results into account.
* Who are willing to sign the informed consent form prior to initiation of any study procedure.

Exclusion Criteria:

Participants who meet any of the following criteria are not eligible for enrollment.

* Who are pregnant or lactating. Women of child bearing potential must avoid becoming pregnant (use of an effective method of contraception or abstinence) for the duration of their participation in the study.
* Who have a known allergy to any component of the Fluzone® Intradermal vaccine, including egg protein, or have had a severe allergic reaction to a previous dose of any influenza vaccine.
* Who have a known or suspected congenital or acquired immunodeficiency or who have had immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months.
* Who have received systemic steroid therapy at any dose or intra-articular administration of steroids within 3 months prior to the day of vaccination.
* Who have received a cumulative dose of inhaled and/or intranasally administered corticosteroids ≥ 880 mcg/day fluticasone equivalent within 3 months prior to the day of vaccination.
* Who have a chronic illness, including but not limited to, cardiac, renal, or auto-immune disorders, or diabetes, at a stage that could interfere with study conduct or completion, based on the opinion of the Investigator.
* Who have a neoplastic disease or any hematologic malignancy, (excluding uncomplicated non-melanoma skin cancer and participants who have a history of neoplastic disease and have been disease free for at least five years).
* Who have participated in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the four weeks preceding the study vaccination or who plan to participate in another clinical trial during the present study period.
* Who have any skin disease other than AD that might compromise the stratum corneum barrier (e.g., bullous disease, psoriasis, cutaneous T cell lymphoma [also called Mycosis Fungoides or Sezary syndrome], dermatitis herpetiformis, Hailey-Hailey, or Darier's disease).
* Who have received blood or blood-derived products that might interfere with the assessment of immune response in the past 3 months prior to vaccination or who plan to receive such products during the study period.
* Who have received previous vaccination (Fluzone® or another vaccine) against influenza in the past 6 months prior to vaccination.
* Who have received any other vaccinations in the 4 weeks preceding study vaccination or who plan to receive any vaccination in the 4 weeks following study vaccination.
* Who have had thrombocytopenia or bleeding disorder in the 3 weeks preceding vaccination.
* Who have had a personal or family history of Guillain-Barré Syndrome.
* Who have a first degree relative already enrolled in the study.
* Who are determined to be not eligible based on the opinion of the Investigator.
* Who require Class I or II topical corticosteroids or calcineurin inhibitors for long-term control of their eczema.

Temporary Vaccination Exclusion Criteria:

Should one of the conditions listed below occur, the Investigator will postpone vaccination until the condition is resolved.

* Signs and symptoms of an acute infectious respiratory illness.
* Febrile illness (temperature ≥ 37.5°C [or ≥ 99.5°F]) or moderate or severe acute illness/infection on the day of vaccination.
* Atopic dermatitis flare, a worsening of the AD participant's skin condition, requiring increased level of baseline treatment during the previous 7 days. Participant must not have applied Class I or II topical corticosteroids or calcineurin inhibitors to any part of the body in the 7 days prior to vaccination. Non-class I or II topical corticosteroids must not have been applied to the deltoid region of the extremity to be vaccinated in the 7 days prior to vaccination.
* Who have taken antipyretics and/or analgesics (e.g. acetaminophen, ibuprofen) within 24 hours prior to the time of vaccination.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-11; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline (Day 0) HAI Antibody Titers | Baseline (Day 0) and Day 28
  The variance of the log fold change from baseline in HAI antibody titers for non-atopic controls and ADEH- participants, following administration per label of a single dose of the seasonal 2011-2012 Fluzone® Intradermal vaccine.

SECONDARY OUTCOMES:
Change from Baseline (Day 0) Influenza-specific T Cell Populations | Baseline (Day 0) and Day 28
  Influenza-specific effector CD4+ and CD8+ T cells pre-vaccination (Day 0) and post-vaccination (Day 28) as measured by flow cytometry for MIP1b, Ki67, CD107a, and CD103 expression.
Change from Baseline (Day 0) Influenza-specific Interferon Gamma and/or Granzyme B Producing Cells | Baseline (Day 0) and Day 28
  Influenza-specific Interferon gamma and/or granzyme B producing cells measured pre-vaccination (Day 0) and post-vaccination (Day 28) by Enzyme-Linked Immunosorbent Spot (ELISPOT).
Change from Baseline (Day 0) Microarray Analysis | Baseline (Day 0), Day 3, and Day 7
  Gene expression profiles of PBMCs pre-vaccination (Day 0) and post-vaccination (Days 3 and 7) as measured by microarray analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Leung, MD, PhD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

REFERENCES:
- [Background] Leung DYM, Jepson B, Beck LA, Hanifin JM, Schneider LC, Paller AS, Monti K, David G, Canniff J, Lorenzo MG, Weinberg A. A clinical trial of intradermal and intramuscular seasonal influenza vaccination in patients with atopic dermatitis. J Allergy Clin Immunol. 2017 May;139(5):1575-1582.e8. doi: 10.1016/j.jaci.2016.12.952. Epub 2017 Feb 13. PMID 28209343
- See also: Atopic Dermatitis Research Network (ADRN) — http://www.nationaljewish.org/adrn/index/
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/